CLINICAL TRIAL: NCT01017796
Title: The Effect of Acetylcysteine and Ascorbic Acid on the Prevention of Radiographic-contrast-agent Induced Reduction in Renal Function in ICU Patients.
Brief Title: Contrast Agent-associated Nephrotoxicity in Intensive Care Unit Patients
Acronym: ICU
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Thessaly (Other)
Responsible Party: Zakynthinos E, Intensive Care Unit department University Hospital Larisa.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KN19201; KIMNEF681264; KIMNEF681264 (Other Grant/Funding Number: UThessaly)
Record Dates: First submitted 2009-11-20; First posted 2009-11-23 (Estimated); Last update posted 2009-11-23 (Estimated); Status verified 2009-11

CONDITIONS: Contrast Induced Nephropathy
Keywords: Contrast induced nephropathy
MeSH Terms: interventions — Acetylcysteine; Ascorbic Acid

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A. Experimental (Experimental): 1200mg acetylcysteine and 2g ascorbic acid at least 2 hours before the start of the index procedure, followed by 1200mg acetylcysteine and 1,5g ascorbic acid the night and the morning after the examination.
  Interventions: Drug: N-acetylcysteine and ascorbic acid
- B. Control (Placebo Comparator): 200ml 0,9% normal saline IV
  Interventions: Drug: N-acetylcysteine and ascorbic acid

INTERVENTIONS:
Drug: N-acetylcysteine and ascorbic acid — 1200mg acetylcysteine and 2g ascorbic acid in 200 ml 0,9% normal saline at least 2 hours before the start of the index procedure, followed by 1200mg acetylcysteine and 1,5g ascorbic acid the night and the morning after the examination.

SUMMARY:
The use of N-acetylcysteine and ascorbic acid reduce the incidence of radiographic contrast agent induced reduction in renal function in Intensive Care Unit patients.

DETAILED DESCRIPTION:
Introduction: Administration of radiographic contrast agents often result in a reversible acute reduction in renal function that begins soon after contrast dye administration.

The incidence of contrast induced nephropathy varies from 5% to 50% depending on the patients' population and the criteria for contrast induced nephropathy (CIN), definition used and it is considered as one of the leading causes of hospital acquired acute renal failure.

The pathogenesis of contrast-induced nephropathy is uncertain. There are two main theories. According to the first one a possible influence on renal hemodynamics, mainly vasoconstriction, resulting in medullary ischemia possibly mediated by an alteration in endothelin and adenosine. In addition to direct vasoconstriction of renal vessels, iodinated contrast agents also block an important pathway for vasodilation and autoregulation possibly by reducing the production of nitric oxide. And according to the other main theory contrast agents exert direct toxic effects on tubular epithelial cells. It seems that reactive oxygen species have a role in CIN.

A lot of studies had examined the incidence of contrast agent-associated nephrotoxicity mainly in stable patients undergoing elective radiographic procedures.

Numerous agents have been examined for their ability to prevent contrast-induced decreases in renal function. Among them the use of low-osmolarity, non anionic contrast agents, and prophylactic hydration have reduced the incidence of CIN. Administration of drugs such as calcium antagonists, theophyllin, dopamine and atrial natriuretic peptide does not prevent CIN. In some studies antioxidant agents like acetylcysteine and ascorbic acid seem to reduce the incidence of CIN.

Critically ill patients represent an absolutely discrete group because they may have acute decrease in renal function, multiple organ failure and they often receive multiple potentially nephrotoxic agents like antibiotics, vasoconstrictives, NSAIDs etc. Critically ill patients frequently required radiographic studies with contrast agent administration in order to improve diagnostic accuracy in the detection of abscesses, or in the diagnosis of suspected embolism. Radiographic studies are often done on an emergent or urgent basis so there is not enough time for patients to receive prophylactic regiments. Despite improvements in supportive care, acute renal failure increases the morbidity and mortality rates in critically ill patients.

We think that it is important initially to investigate the incidence of CIN in critically ill patients a fact that is not established (there is only one retrospective cohort study) and after that to see the impact of a combination of prophylactic strategies in this population.

The ability to prevent CIN in high risk patients will result in significant public health benefits by reducing in-hospital mortality, the hospital stay and the need for dialysis and subsequent the devastating cost of hospitalization.

N-acetylcysteine is a reduced thiol, which is a potent antioxidant that may scavenge a wide variety of oxygen derived free radicals. Ascorbic acid is a potent antioxidant capable of scavenging a wide array of reactive oxygen species and additionally it can regenerate other antioxidants. Acetylcysteine and ascorbic acid are inexpensive treatments with generally mild adverse effects.

Material and methods: This study represent a prospective randomized open label controlled trial. The study will take place in the intensive care unit of the University Hospital of Larissa. Consecutive sampling will be used to recruit patients hospitalized in the ICU department between October of 2009 and October of 2010. The patients who undergo radiographic studies with the administration of contrast agent will be randomly assigned to receive IV either 1200mg acetylcysteine and 2g ascorbic acid or placebo at least 2 hours before the start of the index procedure, followed by 1200mg acetylcysteine and 1,5g ascorbic acid or placebo the night and the morning after the examination. All the patients independently from the randomization will receive hydration with at least 100ml/h IV 0,9% or 0,45% sodium chloride in water, from randomization until at least 6 hours after the examination. The variation of the hydration type and rate allowed for adjustment according the special needs of every patient.

An acute contrast induced reduction in renal function was defined as an increase in the serum creatinine concentration of at least 0,5mg/dl at 72 hours after the injection of the radiocontrast medium or a relative rise of at least 25% fro baseline.

Baseline serum creatinine and urea concentration will be measured from blood sample drawn at the time of randomization, and the follow-up serum urea and creatinine concentration will be measured the 1st, the 2nd and 3rd day after the examination. At the same time intervals we will study the renal function using more sensitive tests like serum cystatin and serum lipocalin (NGAL).

We also will examine the plasma total antioxidant status from blood and urine samples drawn at the time of randomization at the beginning of the procedure and during the following morning.

The daily urine output will also be registered the day before the study and the three subsequent days.

Authorization has been given from the Scientific Council and the Ethical Committee of our hospital.

Clinical and biochemical characteristics of the study patients will include demographic data, diagnosis on admission in ICU, APACHE II score on admission and before randomization, medical history as the presence of cardiac insufficiency, hypertension, coronary disease, hepatic insufficiency, diabetes mellitus, hyperlipidemia, nephrotoxic medications which patients receive like antibiotics, NSAID, chemotherapeutic agents, diuretics, inotropic and vasopressor agents, ACE inhibitors, calcium antagonists,mechanical ventilation during ICU, ICU length of stay, and ICU outcome, the need for renal replacement therapy, the quantity of received radiocontrast agent and the route of administration.

Statistical analysis. All analysis will be performed on an intention-to-treat basis and probability values will be 2-sided. Data will presented as mean +/- SD and 95% CI for continuous variables and as percentage for discrete variables. Analysis will performed using statistical software, SISS 15 for Windows. Data will be compared between the two groups. Characteristics will be compared using the x2 test and the t-test.

ELIGIBILITY:
Inclusion Criteria:

* Presence in the Intensive Care Unit
* Patients undergoing radiologic examinations with the use of IV contrast agents.

Exclusion Criteria:

* Renal failure under renal replacement therapy
* Unstable renal function ( change of serum creatinine between two subsequent days greater than 20% at least 3 days before the study)
* IV administration of contrast agent within the previous 6 days from the study
* Use of ascorbic acid or acetylcysteine during the week before the study
* Pregnancy

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2009-01; Primary Completion 2010-01 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
Morbidity in the Intensive Care Unit | 1,5 year

SECONDARY OUTCOMES:
Incidence of acute nephropathy after administration of radiocontrast agents | 1,5 year

REFERENCES:
- [Derived] Palli E, Makris D, Papanikolaou J, Garoufalis G, Tsilioni I, Zygoulis P, Zakynthinos E. The impact of N-acetylcysteine and ascorbic acid in contrast-induced nephropathy in critical care patients: an open-label randomized controlled study. Crit Care. 2017 Oct 31;21(1):269. doi: 10.1186/s13054-017-1862-3. PMID 29089038